CLINICAL TRIAL: NCT03410641
Title: The Effect of Lifestyle Intervention on the Risk of Cancer - A Study of Participants in the Oslo Diet and Antismoking Study
Brief Title: Long-term Cancer Risk in the Randomised Oslo Diet and Antismoking Study
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Paula Berstad, Principal Investigator, Oslo University Hospital
Other Study IDs: 2016/1442
Record Dates: First submitted 2018-01-08; First posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Cancer; Gastrointestinal Cancer; Lung Cancer; Urinary Tract Cancer; Prostate Cancer
Keywords: cancer risk; randomised trial; intervention; smoking cessation; dietary intervention; weight loss
MeSH Terms: conditions — Neoplasms; Gastrointestinal Neoplasms; Lung Neoplasms; Urologic Neoplasms; Prostatic Neoplasms; Smoking Cessation; Weight Loss | interventions — Diet

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diet and antismoking advice: Dietary and antismoking advice, aiming to reduce participant's risk of cardiovascular diseases
  Interventions: Behavioral: Diet and antismoking advice
- Control: No intervention

INTERVENTIONS:
Behavioral: Diet and antismoking advice — Dietary advice with the aim of reducing participant's serum cholesterol levels, including reduction in the intake of saturated fat and cholesterol, and increased intake of polyunsaturated fat, fish, vegetables and fruit. Weight reduction was recommended for overweight men, as well as reduced consumption of sugar rich foods and drinks, and alcoholic beverages. Smokers were advised to stop smoking. The advice was given both individually and in group sessions during a five-year time period from 1972/3 until 1977/8.
  Groups: Diet and antismoking advice

SUMMARY:
This study examines the effect of a five-year multifactorial lifestyle intervention in the Oslo diet and antismoking study on long-term cancer risk. In 1972-1973, 1232 men with high cardiovascular risk profile were randomised to intervention including cholesterol lowering diet, weight loss and antismoking advice, or control (1:1). This study examines the effect of the intervention on 43-year cancer incidence and mortality.

DETAILED DESCRIPTION:
The Oslo diet and antismoking study showed that a 5-year lifestyle intervention reduced the long-term risk of coronary events and mortality. The lifestyle risk factors for cancer are partly similar to those for coronary heart disease, e.g. smoking, high body weight, unfavourable diet. The investigators therefore expect that the intervention has an effect on cancer risk in the long term.

In this follow-up study, the investigators analyse the association between the intervention, and cancer incidence and mortality drawn from the Cancer Registry of Norway and the Norwegian Cause of Death Registry from the time of randomisation in 1972/3 until the end of 2015.

ELIGIBILITY:
Inclusion Criteria:

* participated in screening of coronary risk factors, into which all men born in 1923-1932 and living in Oslo were invited in 1972-1973
* being in the upper quartile of a coronary risk score based on blood pressure, serum total cholesterol concentration and cigarette smoking

Exclusion Criteria:

* serum total cholesterol level above 9.0 mmol per Liter
* having a healthy diet, based on a short dietary history
* self-reported cardiovascular disease or diabetes
* previous history of cancer

Ages: 40 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants selected for this follow-up study (n=1216) are the eligible subjects of the 1232 men at high cardiovascular risk profile who participated in the Oslo Diet and Antismoking Study (included in 1972-73). Fourteen men were excluded because they did not consent to studies other than the main study, and two more because of previous history of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1216 (Actual)
Dates: Start 1972-01-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of the group of cancers related to smoking, diet or body mass index | 43 years
  Diagnosis of carcinoma in the oral cavity, oropharynx, esophagus, stomach, colorectum, liver and intrahepatic bile ducts, pancreas, larynx, trachea, bronchus and lung, urinary tract and thyroid gland, drawn from the Cancer Registry of Norway

SECONDARY OUTCOMES:
Mortality in the group of cancers related to smoking, diet or body mass index | 43 years
  Mortality in cancers in the oral cavity, oropharynx, esophagus, stomach, colorectum, liver and intrahepatic bile ducts, pancreas, larynx, trachea, bronchus and lung, urinary tract and thyroid gland, drawn from the Norwegian Cause of Death Registry
Cancer incidence | 43 years
  Any cancer diagnosis, drawn from the Cancer Registry of Norway
Cancer mortality | 43 years
  Mortality in any cancer, drawn from the Norwegian Cause of Death Registry
Incidence of gastrointestinal cancer | 43 years
  Diagnosis of carcinoma in gastro-intestinal tract, drawn from the Cancer Registry of Norway
Incidence of lung cancer | 43 years
  Diagnosis of carcinoma in lung, drawn from the Cancer Registry of Norway
Incidence of urinary tract cancer | 43 years
  Diagnosis of carcinoma in urinary tract, drawn from the Cancer Registry of Norway
Incidence of prostate cancer | 43 years
  Diagnosis of carcinoma in prostate, drawn from the Cancer Registry of Norway

CONTACTS AND LOCATIONS:
Overall Officials: Paula Berstad, PhD, Principal Investigator — Norwegian Institute of Public Health

IPD SHARING:
Plan to Share IPD: No